CLINICAL TRIAL: NCT02523612
Title: Prospective National Multicentre Study to Validate a Model of Surgical Deescalation in Atypicals Breast Lesions
Brief Title: Study to Validate a Model of Surgical Deescalation in Atypicals Breast Lesions
Acronym: NOMAT01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-A00045-44; 2015/2211 (Other: CSET number)
Record Dates: First submitted 2015-08-06; First posted 2015-08-14 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with atypical lesions (Experimental)
  Interventions: Procedure: Biopsy; Procedure: Blood sample

INTERVENTIONS:
Procedure: Biopsy
Procedure: Blood sample

SUMMARY:
Routine screening mammography has increased the non-palpable suspicious lesion detection rate, requiring histopathological evaluation. The discovery of atypical lesions on the breast biopsy is associated with two interrelated risks:

1. The risk of underestimating the severity of the lesion biopsied currently leads systematically to achieve a surgical resection for these patients while a breast cancer (BC) will finally identified at surgery in 10 to 25% of cases. Thus, unnecessary surgeries will be performed in 75 to 90% of cases (no cancer).
2. These breast lesions confer long-term increase in the subsequent risk of breast cancer (cumulative incidence of 15 to 25% at 25 years). Thus, women identified with atypical lesions are then followed using clinical and mammographic annual evaluation.

The goal would be to get a model to assess the risk and no longer operate those patients at high risk of BC. Several groups have attempted to identify predictors of concurrent or secondary BC associated with the discovery of an unusual lesion at biopsy. However, they are often focused on a subtype of atypia (eg atypical metaplasia, atypical ductal hyperplasia, atypical lobular hyperplasia) and no prediction model has been validated in prospective multicenter. Based on a large retrospective study at Gustave Roussy, a prediction model (Nomat) has been developed, common to all atypical lesions, which can predict the presence of a BC at excision surgery (risk of concurrent BC). This model is based on the age of the patient, the disappearance of radiographic abnormalities (microcalcifications in general) after the biopsy and initial radiological lesion size. This model has good performance with an area under the curve (AUC) of 0.72. In previous series, with a BC high-risk threshold of 20%, negative predictive value was 90%, and this model would have prevented the surgery in 51% of patients (low risk patients by model). It is essential to validate this model by forward-looking and in different centers to ensure its relevance.

This is a multicenter prospective validation of the model on 300 patients operated for atypical lesions in 21 centers. All patients with atypical breast lesions have a routine surgery. The clinical data, imaging and histological data will be collected prospectively. The main objective of this study is to validate the model Nomat.

ELIGIBILITY:
Inclusion Criteria:

* Women who have had a recent diagnosis of atypical breast lesions (atypical metaplasia, atypical ductal hyperplasia, atypical lobular hyperplasia, lobular carcinoma in situ) on a breast biopsy for microcalcifications on mammography Or for little suspect distortion in ultrasound or mammary MRI.
* Report of the anatomopathological examination of the biopsy allowing the diagnosis of an atypical lesion available
* Patient 18 years or more
* Informed consent signed.
* Patient affiliated to a system of social security or beneficiary of such plan
* General condition ECOG-OMS 0 or 1

Exclusion Criteria:

* Nodular lesion associated with ultrasound or mammography opacity
* Palpable nodule
* Presence of ductal carcinoma in situ or invasive carcinoma associated to biopsy
* Personal history of breast cancer or homo contralateral
* Previous history of breast irradiation or breast cancer or other area for malignancy (Hodgkin, etc ...)
* Women with a BRCA1 or BRCA2 mutation diagnosed or other genetic predisposition to breast cancer and highly penetrant autosomal dominant.
* Pregnant or nursing women
* Women with a cons-indication or refusal of surgery
* Private Women of freedom under guardianship.
* Presence of aggressive lobular in situ carcinoma (pléioforme, Florida or necrosis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-06-24 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Negative Predictive value of the NOMAT model | Up to 3 months
  The primary endpoint is the negative predictive value (NPV) of Nomat model used to predict the absence of breast cancer associated with cases of atypical lesions in breast biopsy

SECONDARY OUTCOMES:
Exploratory research for biomarkers using DNA Seq | Up to 3 months
  The study will be Nomat parallel homogeneous database of prospective clinical and pathological data of patients operated for atypical breast lesions associated with tissue and blood samples (5 mL in EDTA tube).
  This bank will exploratory research of new biomarkers and validation of new biomarkers that may emerge in the coming years.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Uzan C, Mazouni C, Rossoni C, De Korvin B, de Lara CT, Cohen M, Chabbert N, Zilberman S, Boussion V, Vincent Salomon A, Espie M, Coutant C, Marchal F, Salviat F, Boulanger L, Doutriaux-Dumoulin I, Jouve E, Mathelin C, de Saint Hilaire P, Mollard J, Balleyguier C, Joyon N, Triki ML, Delaloge S, Michiels S. Prospective Multicenter Study Validate a Prediction Model for Surgery Uptake Among Women with Atypical Breast Lesions. Ann Surg Oncol. 2021 Apr;28(4):2138-2145. doi: 10.1245/s10434-020-09107-z. Epub 2020 Sep 12. PMID 32920723